CLINICAL TRIAL: NCT06767293
Title: I-InTERACT Preterm Parenting Randomized Controlled Trial
Brief Title: I-InTERACT Preterm Parenting
Acronym: I2P-RCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024-0349
Record Dates: First submitted 2024-11-12; First posted 2025-01-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Child Behavior Problem; Preterm; Parent-Child Relations; Parenting
Keywords: telehealth; online learning; microlearning
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Masking for outcomes assessor for DPICS study measure
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- I-InTERACT Intervention (I2P) with regularly scheduled therapist coaching (Active Comparator)
  Interventions: Behavioral: I-InTERACT Parenting Intervention (I2P) and coaching sessions
- I-InTERACT Microlearning Intervention (I2P-Micro) with regularly scheduled therapist coaching (Active Comparator)
  Interventions: Behavioral: I-InTERACT Parenting Microlearning Intervention (I2P Micro) and coaching sessions
- Internet Resource Group (Other): Control condition
  Interventions: Other: Internet Resources

INTERVENTIONS:
Behavioral: I-InTERACT Parenting Intervention (I2P) and coaching sessions — Online learning sessions for parents of preterm children
  Arms: I-InTERACT Intervention (I2P) with regularly scheduled therapist coaching
Behavioral: I-InTERACT Parenting Microlearning Intervention (I2P Micro) and coaching sessions — Online microlearning sessions for parents of preterm children
  Arms: I-InTERACT Microlearning Intervention (I2P-Micro) with regularly scheduled therapist coaching
Other: Internet Resources — control condition
  Arms: Internet Resource Group

SUMMARY:
Many children born very preterm experience behavior problems, and existing resources for parenting these children are lacking. A pilot trial established the effectiveness of a preterm parenting intervention, I-Interact Preterm (I2P). This study proposes a three-arm randomized controlled trial (RCT) comparing the established seven-session I2P program, a microlearning delivery mode (I2P-Micro), and an internet resource comparison group (IRC). Outcomes will be assessed at pretreatment, post-treatment (12 weeks later), and at an extended follow-up six months post-randomization. These outcomes include parenting behaviors, child behavior problems, and parent distress. It is anticipated that both I2P and I2P-Micro will result in significant improvements relative to the IRC condition, with greater utilization expected in the I2P-Micro group.

DETAILED DESCRIPTION:
Many children born very preterm or extremely preterm exhibit a distinct behavioral phenotype characterized by impairments in cognition and attention and concomitant social and emotional problems. These children are significantly more likely to develop ADHD than children born at term and have similar rates of comorbid symptoms such as noncompliance, emotionality, and attention-seeking behaviors as those observed in children with ADHD. Although addressing children's mental health and behavioral challenges is a priority identified by parents, evidence-based interventions to promote effective parenting and mitigate child behavior problems in this population are lacking.

From 2021-2022, a single-arm pilot clinical trial was conducted for children born very preterm using content adapted from previous trials of I-InTERACT North and I-InTERACT Express, which included seven sessions and weekly online coaching from a therapist. Children demonstrated a significant reduction in externalizing behavior problems from pre- to post-intervention, and caregivers' positive parenting skills significantly increased during the same period.

Given relatively high rates of attrition in the pilot trial and stakeholder feedback regarding challenges in completing the program, the utility of microlearning delivery-delivering content in approximately 5-minute segments-will be tested relative to the existing I-InTERACT Preterm program and an internet resource comparison group. This approach is anticipated to improve uptake, engagement, and retention, particularly for young adults who routinely consume information in this format, while maintaining the efficacy of the original program.

A three-arm randomized controlled trial (RCT) is proposed to compare the seven-session I2P program to the microlearning delivery mode (I2P-Micro) and an internet resource comparison group (IRC). Participants in the I2P and I2P-Micro groups will also meet weekly or biweekly with a trained therapist to review content and receive coaching while practicing skills. Outcomes will be assessed at pretreatment, post-treatment (12 weeks later), and at an extended follow-up six months post-randomization. These outcomes include parenting behaviors, child behavior problems, and parent distress. It is anticipated that both I2P and I2P-Micro will result in significant improvements relative to the IRC condition, with greater utilization expected in the I2P-Micro group.

ELIGIBILITY:
Inclusion Criteria:

* Born at < 32 weeks gestational age.
* Total T score of > 55 on the Child Behavior Checklist Total or Externalizing Behavior Scales OR Total T score of > 55 on the Eyberg Child Behavior Inventory total problem- or total intensity-scale.
* English is the primary spoken language in the home.

Exclusion Criteria:

* Is not 18 years or older.
* Participant will be excluded from the study if the child does not reside with the caregiver at least half-time; the caregiving situation is not stable (i.e., there must be no scheduled custody hearings).
* English is not the primary language spoken in the home.
* Caregivers with a psychiatric hospitalization in the past year.

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2024-11-27 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Dyadic Parent-Child Interaction Coding System Total Positive Parenting Behavior Score | 3 months post baseline and 6 months post baseline
  Minimum score is 0, maximum score is not applicable as parents may exhibit any number of positive behaviors during the time frame data is collected. A higher score means a greater number of positive parenting behaviors were exhibited, which is considered better.
Child Behavior Checklist Externalizing T-score | 3 months post baseline and 6 months post baseline
  Minimum t score for girls is 33, and maximum t score is 100. Minimum t score for boys is 34 and maximum t score is 100. A higher t score indicates more externalizing behaviors, which is considered worse.

SECONDARY OUTCOMES:
ECBI Intensity T-Score | 3 months post baseline and 6 months post baseline
  The ECBI Problem T-Score is a 36-item checklist of concerns (e.g., noncompliance, emotionality, attention-seeking) will be used to assess the number and intensity of child behavior problems pre- and post-treatment. On the ECBI, the parent rates how often each behavior occurs (7-point intensity scale), and whether the behavior is a problem (Yes/No Problem Scale). Higher T-Scores indicate greater intensity of problem behaviors. The lowest T-Score is 36 and the highest is 252, with a clinical cut-off at 60. During screening for this study, a T-Score greater than 55 for this scale meets meeting eligibility criteria.
ECBI Problem T-Score | 3 months post baseline and 6 months post baseline
  The ECBI Problem T-Score is a 36-item checklist of concerns (e.g., noncompliance, emotionality, attention-seeking) will be used to assess the number and intensity of child behavior problems pre- and post-treatment. On the ECBI, the parent rates how often each behavior occurs (7-point intensity scale), and whether the behavior is a problem (Yes/No Problem Scale). Higher T-Scores indicate more challenging behaviors. The lowest T-Score is 41 and the highest is 88, with a clinical cut-off at 60. During screening for this study, a T-Score greater than 55 for this scale meets meeting eligibility criteria.
Caregiver Psychological Distress | 3 months post baseline and 6 months post baseline
  Caregiver psychological distress will be assessed using the CES-D, a 20-item self-report inventory in which participants rate how often over the last week they have been bothered by various symptoms of depression in the last week. Total scores range from 0 to 60, with higher scores indicate greater caregiver distress. Scores 16 and above indicate a risk for clinical depression.

OTHER OUTCOMES:
Parental Stress | 3 months post baseline and 6 months post baseline
  The Parental Stress Scale attempts to measure the levels of stress experienced by parents through an 18-item self-report measure. Questions are answered on a 5-Point Likert scale. Higher scores indicate a higher level of parental stress. There are no clinical cut-offs.
Positive Attitude Towards Child | 3 months post baseline and 6 months post baseline
  Positive attitude towards the child will be measured using the Five-Minute Speech Sample (FMSS), which is a procedure designed to assess expressed emotion in caregivers by asking respondents to talk for five uninterrupted minutes about their thoughts and feelings about a subject and how they get along together. The speech sample is coded, with a greater number of positive responses coded indicating a greater positive attitude towards their child.

CONTACTS AND LOCATIONS:
Overall Officials: Shari Wade, PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
Only de-identified data will be shared.

REFERENCES:
- [Background] Ask H, Gustavson K, Ystrom E, Havdahl KA, Tesli M, Askeland RB, Reichborn-Kjennerud T. Association of Gestational Age at Birth With Symptoms of Attention-Deficit/Hyperactivity Disorder in Children. JAMA Pediatr. 2018 Aug 1;172(8):749-756. doi: 10.1001/jamapediatrics.2018.1315. PMID 29946656
- [Background] de Silva A, Neel ML, Maitre N, Busch T, Taylor HG. Resilience and vulnerability in very preterm 4-year-olds. Clin Neuropsychol. 2021 Jul;35(5):904-924. doi: 10.1080/13854046.2020.1817565. Epub 2020 Sep 13. PMID 32924801
- [Background] Jones K, Daley D, Hutchings J, Bywater T, Eames C. Efficacy of the Incredible Years Programme as an early intervention for children with conduct problems and ADHD: long-term follow-up. Child Care Health Dev. 2008 May;34(3):380-90. doi: 10.1111/j.1365-2214.2008.00817.x. PMID 18410644
- [Background] Williams TS, McDonald KP, Roberts SD, Westmacott R, Dlamini N, Tam EWY. Understanding Early Childhood Resilience Following Neonatal Brain Injury From Parents' Perspectives Using a Mixed-Method Design. J Int Neuropsychol Soc. 2019 Apr;25(4):390-402. doi: 10.1017/S1355617719000079. PMID 31050330
- [Background] Wang C, Bakhet M, Roberts D, Gnani S, El-Osta A. The efficacy of microlearning in improving self-care capability: a systematic review of the literature. Public Health. 2020 Sep;186:286-296. doi: 10.1016/j.puhe.2020.07.007. Epub 2020 Aug 31. PMID 32882481
- [Background] De Gagne JC, Woodward A, Park HK, Sun H, Yamane SS. Microlearning in health professions education: a scoping review protocol. JBI Database System Rev Implement Rep. 2019 Jun;17(6):1018-1025. doi: 10.11124/JBISRIR-2017-003884. PMID 30489350